CLINICAL TRIAL: NCT00371280
Title: Prosthetic Motility and Complications in Pegged Versus Unpegged Hydroxyapatite Orbital Implants
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8422
Record Dates: First submitted 2006-09-01; First posted 2006-09-04 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2008-06

CONDITIONS: Anophthalmos; Orbital Implants
Keywords: hydroxyapatite; peg; prosthetic motility; orbital implant
MeSH Terms: conditions — Anophthalmos | interventions — Orbital Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Pegged unpegged hydroxyapatite orbital implantation
  Interventions: Procedure: orbital implant
- 2 (Active Comparator): Unpegged hydroxyapatite orbital implantation
  Interventions: Procedure: orbital implant

INTERVENTIONS:
Procedure: orbital implant — Implantation of pegged versus unpegged hydroxyapatite orbital implants

SUMMARY:
Pegging the hydroxyapatite for increasing prosthetic motility sometimes leads to some complications for the patient. These complications ranging from discharge, granuloma formation, exposure, implant infection to socket discomfort and etc. We are going to compare prosthetic motility, objectively and subjectively (patients satisfaction) before and after pegging the hydroxy- apatite, and evaluate the complications after pegging.

ELIGIBILITY:
Inclusion Criteria:

* orbital hydroxyapatite implants

Exclusion Criteria:

* history of systemic disease
* history of radio therapy
* secondary hydroxapatite implant
* complications lead to re-surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-11; Primary Completion 2006-10 (Estimated); Study Completion 2006-11 (Estimated)

PRIMARY OUTCOMES:
Changing movement in up gaze: 0.58 mm
Changing movement in down gaze: 0.83 mm
Changing movement in medial gaze: 0.75 mm
Changing movement in lateral gaze: 1.2 mm

CONTACTS AND LOCATIONS:
Overall Officials: Babak Babsharif, MD, Principal Investigator — Ophthalmic Research Center of Shaheed Beheshti Medical University
Locations (1):
- Babak Babsharif, MD, Tehran, Tehran Province, Iran